CLINICAL TRIAL: NCT03335020
Title: Assessment of Contrast-enhanced Ultrasonography, Shear Wave Elastography, Strain Imaging, and 3-D Volume Ultrasonography on Arterial Wall Visualization and Stiffness in Patients With Fibromuscular Dysplasia...
Brief Title: Using Ultrasonography, Shear Wave Elastography, Strain Imaging, and 3-D Volume Ultrasonography on Cardiovascular Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed by Investigator
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew W. Urban, Associate Professor of Biomedical Engineering, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-000020
Record Dates: First submitted 2017-10-04; First posted 2017-11-07 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Fibromuscular Dysplasia of Arteries; Segmental Arterial Mediolysis; Spontaneous Coronary Artery Dissection; Atherosclerosis of Artery
Keywords: Ultrasound; 3D ultrasonography; Contrast-enhanced ultrasound; Shear wave elastography
MeSH Terms: conditions — Fibromuscular Dysplasia; Coronary Artery Dissection, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Normal (Placebo Comparator): Healthy volunteers. Assessment using Shear Wave Elastography, Pulse Wave Imaging, Contrast-Enhanced Ultrasound, Strain Imaging and 3-D Volume ultrasound
  Interventions: Device: Shear Wave Elastography; Device: Pulse Wave Imaging; Drug: Contrast-Enhanced Ultrasound; Other: Strain Imaging; Device: 3-D Volume Ultrasound
- Fibromuscular Dysplasia (FMD) (Active Comparator): Subjects with diagnosis of FMD. Assessment using Shear Wave Elastography, Pulse Wave Imaging, Contrast-Enhanced Ultrasound, Strain Imaging and 3-D Volume ultrasound
  Interventions: Device: Shear Wave Elastography; Device: Pulse Wave Imaging; Drug: Contrast-Enhanced Ultrasound; Other: Strain Imaging; Device: 3-D Volume Ultrasound
- Atherosclerosis (Active Comparator): Subjects with diagnosis of atherosclerosis. Assessment using Shear Wave Elastography, Pulse Wave Imaging, Contrast-Enhanced Ultrasound, Strain Imaging and 3-D Volume ultrasound
  Interventions: Device: Shear Wave Elastography; Device: Pulse Wave Imaging; Drug: Contrast-Enhanced Ultrasound; Other: Strain Imaging; Device: 3-D Volume Ultrasound
- Spontaneous Coronary Artery Dissection (SCAD) (Active Comparator): Subjects with diagnosis of SCAD. Assessment using Shear Wave Elastography, Pulse Wave Imaging, Contrast-Enhanced Ultrasound, Strain Imaging and 3-D Volume ultrasound
  Interventions: Device: Shear Wave Elastography; Device: Pulse Wave Imaging; Drug: Contrast-Enhanced Ultrasound; Other: Strain Imaging; Device: 3-D Volume Ultrasound
- Segmental Arterial Mediolysis (SAM) (Active Comparator): Subjects with diagnosis of SAM. Assessment using Shear Wave Elastography, Pulse Wave Imaging, Contrast-Enhanced Ultrasound, Strain Imaging and 3-D Volume ultrasound
  Interventions: Device: Shear Wave Elastography; Device: Pulse Wave Imaging; Drug: Contrast-Enhanced Ultrasound; Other: Strain Imaging; Device: 3-D Volume Ultrasound

INTERVENTIONS:
Device: Shear Wave Elastography — The subject will be asked to lay on a hospital bed for ultrasound imaging of the arteries. The subject will have an automatic blood pressure cuff put on to measure blood pressure. The subject will also have a three-lead ECG taken during the experiment. The artery will be visualized using ultrasound imaging, and the depth of the arterial wall will be noted. The focal depth on the device will be set to measure shear wave propagation in the walls of the artery. Measurements will be made at multiple locations along the artery's length and at different phases of the cardiac cycle determined by ECG gating. Either or both the Verasonics or GE Logiq systems will be used for measurements. Measurements made with these systems use acoustic output within the FDA regulatory limits of diagnostic imaging.
  Other Names: Verasonics
Device: Pulse Wave Imaging — Researchers will use the Verasonics device to acquire data for measurement of wave velocity in the tissue of interest (arterial walls and surrounding tissue) due to the pressure pulse from ejection of blood by the heart into the systemic circulation. Using ECG gating we can regulate the timing of the individual acquisitions. In each acquisition, high frame rate ultrasound imaging is used to acquire data to measure the motion of the propagating waves. Multiple measurements on different heartbeats are made with varying delays to obtain measurements throughout the heart cycle assuming at that the behavior during consecutive heartbeats is similar. Multiple measurements will be made in a given artery and multiple locations in the arterial wall.
  Other Names: Verasonics
Drug: Contrast-Enhanced Ultrasound — Will be done using Lumason (Bracco Diagnostics, Inc) administered intravenously via slow hand infusion. Real-time contrast-enhanced carotid cine-loop (longitudinal and short axis) images obtained at least 3 seconds before and 5 minutes after the appearance of the contrast effect in the lumen of the determined artery will be acquired and digitally stored for off line analysis. Up to two vials will be used for a study.
  Other Names: Lumason
Other: Strain Imaging — Measurements will be performed offline on the workstation using Echo PAC software (GE Healthcare Inc., Princeton, NJ). The media-adventitia interface of the arterial wall will be manually traced from a still frame image. The circumferential and radial strain curves will be automatically obtained. Measurements of the peak radial and circumferential strain, strain rate will be obtained. If arterial plaque is identified: A region of interest will be placed at the plaque in 3 different regions: 2 shoulder regions and the fibrous cap top, the measurement results of the peak longitudinal, radial and circumferential strain, strain rate will be acquired by the software.
Device: 3-D Volume Ultrasound — When generating a 3D volume the ultrasound data can be collected in 4 common ways. Freehand, which involves tilting the probe and capturing a series of ultrasound images and recording the transducer orientation for each slice. Mechanically, where the internal linear probe tilt is handled by a motor inside the probe. Using an endoprobe, which generates the volume by inserting a probe and then removing the transducer in a controlled manner. The fourth technology is the matrix array transducer that uses beam steering to sample points throughout a pyramid shaped volume

SUMMARY:
The researchers are trying to see whether contrast-enhanced ultrasonography, shear wave elastography, strain imaging, and 3-D volume ultrasonography improves arterial wall visualization and identifies arterial elastic properties among individuals with fibromuscular dysplasia (FMD), atherosclerosis, personal history of spontaneous coronary artery dissections (SCAD), or personal history of segmental arterial mediolysis (SAM) that may be different compared to those without the aforementioned conditions.

DETAILED DESCRIPTION:
Aims, purpose, or objectives:

1. To describe whether contrast-enhanced ultrasonography, strain imaging, and 3-D volume ultrasonography are helpful to characterize affected arteries and improve the imaging of arterial wall among patients with Fibromuscular Dysplasia (FMD) and segmental arterial mediolysis (SAM).
2. Evaluate the arterial elastic properties of individuals with FMD and compare to normal individuals, those with atherosclerosis disease, those with personal history of spontaneous coronary artery dissections (SCAD), and/or personal history of segmental arterial mediolysis (SAM) by elastography.
3. Identification of vulnerable arterial elastic properties using contrast-enhanced ultrasonography, shear wave elastography, strain imaging, and 3-D volume ultrasonography to predict short-term and long-term outcomes among individuals with FMD, normal individuals, those with atherosclerosis disease, those with SCAD, and/or SAM.
4. Develop risk factor profiles and risk score systems of patients undergoing contrast-enhanced ultrasonography, shear wave elastography, strain imaging, and 3-D volume ultrasonography among individuals with FMD, those with atherosclerosis disease, those with personal history of SCAD, and/or personal history of SAM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromuscular dysplasia (FMD), and/or segmental arterial mediolysis (SAM), and/or spontaneous coronary artery dissection (SCAD), and those with atherosclerosis, and normal individuals.
* Adult male and non-pregnant female patient 18-100 years of age.
* Patients who are able and willing to sign the informed consent will be enrolled.

Exclusion Criteria:

* Missing records to determine whether or not they have fibromuscular dysplasia (FMD), and/or segmental arterial mediolysis (SAM), and/or spontaneous coronary artery dissection (SCAD), and those with atherosclerosis, and normal individuals.
* Patients who do not accept to participate in research studies.
* Prior contraindication to contrast agent.
* Women who are breastfeeding or pregnant
* Patients less than 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects who Completed All of the Ultrasound Examinations | 2 years after starting enrollment
  Completion of ultrasound examinations to determine visualization of arterial wall (contrast-enhanced ultrasound, 3-D volume ultrasound) and its mechanical properties (shear wave elastography, pulse wave imaging, strain imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Urban, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials